CLINICAL TRIAL: NCT01447082
Title: Epidemiology Study to Assess the Safety of a New Slow-release Form of Seroquel (Quetiapine) in the Post-marketing Phase in the UK
Brief Title: General Practice Research Database Seroquel XR Safety Study
Acronym: GPRD SeroquelS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: D1444C00006
Record Dates: First submitted 2011-09-19; First posted 2011-10-05 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Schizophrenia; Major Depressive Disorder; Bipolar Disorder
Keywords: atypical; antipsychotics; quetiapine
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Bipolar Disorder

STUDY DESIGN:
Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Quetiapine XR group
- Non-quetiapine comparison group

SUMMARY:
The main objective of this observational study is to characterize new users of quetiapine XR as well as new users of other study drugs (i.e. the comparison group) and to quantify the risk of developing newly diagnosed outcomes of interest in new users of quetiapine XR as well as in other study drugs.

DETAILED DESCRIPTION:
Epidemiology study to assess the safety of a new slow-release form of Seroquel (quetiapine) in the post-marketing phase in the UK.

ELIGIBILITY:
Inclusion Criteria:

* Episodes of new use (>/=1 prescription) of quetiapine XR or other study drugs

Exclusion Criteria:

* Less than two years of recorded history before the start of the marketing of quetiapine XR (or cohort entry date)
* If the duration and dose of the antipsychotic drug cannot be determined

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of the general population in the UK consisting of 3 millions inhabitants.
Sampling Method: Non-Probability Sample
Enrollment: 37372 (Actual)
Dates: Start 2008-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The outcome of interest will be evaluated by means of relative risk based on incidence rates estimates in users of quetiapine XR vs corresponding incidence rates in users of comparison drugs | During follow-up of a treatment episode estimated to be on average of 1.5 years
Duration of treatment | During follow-up estimated to be on average of 1.5 years.
Duration of treatment episode | During follow-up estimated to be on average of 1.5 years
  Episode, defined as the treatment time from first to last prescription of quetiapine XR or other study drugs.
Comorbidities defined by clinical diagnosis or prescription | Baseline and during follow up of treatment estimated to be on average 1.5 years
Age | Baseline
Gender | Baseline
Dose | During follow-up of treatment estimated to be on average 1.5 years
Adherence | During follow-up of treatment estimated to be on average 1.5 years
The number of subjects to whom the drug was prescribed by the general practitioners. | During follow-up of treatment estimated to be on average 1.5 years
  The number of patients, whom the drug was prescribed by the specified type of prescriber (specialist, general practitioner or another type of physician).
Indication for treatment | During follow-up of treatment estimated to be on averaged 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christoph R Meier, PROF DR PHIL, Principal Investigator — University hospital of Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Switzerland